CLINICAL TRIAL: NCT05917470
Title: A Phase 1/2 Study of ONCT-534 in Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Clinical Study of ONCT-534 in Subjects With Metastatic Castration-resistant Prostate Cancer.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Oncternal Therapeutics, Inc. announced on 12 SEP 2024 its decision to discontinue its clinical trials evaluating ONCT-534, its dual action androgen receptor inhibitor for the treatment of patients with metastatic castration resistant cancer.
Sponsor: Oncternal Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONCT-534-101
Record Dates: First submitted 2023-06-07; First posted 2023-06-23 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Level 1: 40mg QD (Experimental): 40mg of single agent ONCT-534 to be administered daily in oral tablets
  Interventions: Drug: ONCT-534
- Dose Level 2: 80mg QD (Experimental): 80mg of single agent ONCT-534 to be administered daily in oral tablets
  Interventions: Drug: ONCT-534
- Dose Level 3: 160mg QD (Experimental): 160mg of single agent ONCT-534 to be administered daily in oral tablets
  Interventions: Drug: ONCT-534
- Dose Level 4: 300mg QD (Experimental): 300mg of single agent ONCT-534 to be administered daily in oral tablets
  Interventions: Drug: ONCT-534
- Dose Level 5: 600mg QD (Experimental): 600mg of single agent ONCT-534 to be administered daily in oral tablets
  Interventions: Drug: ONCT-534
- Dose Level 6: 1200 mg QD (Experimental): 1200mg of single agent ONCT-534 to be administered daily in oral tablets
  Interventions: Drug: ONCT-534
- BID Dose Level 1: 160 mg BID (Experimental): 600mg of single agent ONCT-534 to be administered daily in oral tablets
  Interventions: Drug: ONCT-534
- BID Dose Level 2: 300 mg BID (Experimental): 300mg of single agent ONCT-534 to be administered twice daily in oral tablets
  Interventions: Drug: ONCT-534

INTERVENTIONS:
Drug: ONCT-534 — ONCT-534 is a dual-action androgen receptor inhibitor (DAARI) with a novel mechanism of action that includes inhibition of AR function and degradation of the AR protein mediated by interaction with the N-terminal domain (NTD) of the AR. ONCT-534 has demonstrated preclinical activity in prostate cancer models against both unmutated androgen receptor (AR), and against multiple forms of AR alteration, including those with AR amplification, mutations in the AR ligand binding domain (LBD), and splice variants with loss of the AR LBD.
  Other Names: GTx-534; UT-34

SUMMARY:
A first-in-human clinical trial to test the investigational treatment ONCT-534 in participants with metastatic castration-resistant prostate cancer. The main questions it aims to answer are:

* What are the most tolerable doses of ONCT-534? (Phase 1)
* Does ONCT-534 have anti-tumor activity at tolerable doses? (Phase 2)

This is a dose escalation and expansion study where participants will receive daily oral doses of ONCT-534.

DETAILED DESCRIPTION:
This is a Phase 1/2 multi-center study to investigate the safety, tolerability, and anti-tumor acitivity of ONCT-534 in patients with relapsed or refractory metastatic castration-resistant prostate cancer. The study consists of 2 phases: a Phase 1 Dose Escalation and a Phase 2 Dose Expansion.

* During the dose escalation in Phase 1 a group of participants will be assigned a certain dose level. Once the dose level is considered safe, the next group will be assigned a higher dose level. The dose level may be raised or lowered depending on any safety events that occur throughout Phase 1. There will be approximately 27 participants enrolled in Phase 1. At the end of Phase 1, two dose levels will be chosen to be tested in Phase 2.
* During Phase 2, participants will be randomly assigned to 1 of the 2 dose levels chose in Phase 1. Approximately 16 participants will be enrolled in each of the 2 dose level groups, for a total of 32 participants.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age
* Subject has histologically documented metastatic adenocarcinoma of the prostate confirmed by biopsy without neuroendocrine differentiation or small cell features.
* Subjects has a history of metastatic CRPC.
* Subject has R/R disease following treatment with at least one next-generation AR-signaling inhibitor.
* Subject has at least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria or evaluable bony disease. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
* Subject has an Eastern Cooperative Oncology Group performance status of 0,1 or 2, and life expectancy of ≥ 6 months.
* Subject agrees to take or continue luteinizing hormone-releasing hormone agonist or antagonist therapy or has undergone bilateral orchiectomy.
* At least 2 weeks or five half-lives have elapsed, whichever is earliest, since last systemic therapy, including taxanes or other chemotherapy. At least one month has elapsed since systemic therapy with radionuclide pharmaceutical agents
* Subject has evidence of disease progression on or after their most recent systemic treatment
* Subject has a PSA level ≥ 10 ng/mL, or ≥ 2 ng/mL and ≥ 50% increase from nadir on prior therapy, whichever is lowest.
* Subject has serum testosterone < 50 ng/dL.
* Subject has adequate renal, hepatic, and pulmonary function
* Subject is committed to practice true abstinence, or use a highly effective method of contraception with any female partner of childbearing potential unless documented to be surgically sterile (i.e., vasectomy or bilateral orchiectomy) and to not make semen donations during the study and for 3 months after the last dose of study drug.

Exclusion Criteria:

* Subject has small cell prostate cancer or neuroendocrine disease histology, including mixed histology.
* Subject has metastases to the brain or central nervous system
* Subject is receiving concurrent anti-cancer therapy (including chemotherapy, antibody therapy, immunotherapy, cellular therapy, or other experimental therapies) except for ongoing androgen inhibiting therapy such as luteinizing hormone-releasing hormone (LHRH) agonists. Supportive non-cancer directed therapies such as bisphosphonates or denosumab are allowed.
* Subjects taking a strong inhibitor of CYP3A4 or a substrate of CYP2C9 or CYP2C19
* Subject had major surgery within 30 days prior to start of study drug.
* Subject has current, untreated pathologic long-bone fractures(s), or risk of imminent pathologic fracture(s).
* Subject has current or imminent spinal cord compression.
* Subject has an active seizure disorder or a history of seizure disorder(s).
* Subject has evidence of active human immunodeficiency virus infection, hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Subject has any other serious illness or medical condition that would interfere with study participation
* Subject has abnormal electrocardiograms (ECGs) that are clinically significant, including average QTcF > 450 ms, or a history of Torsade de Pointes.
* Subject has any infection requiring parenteral antibiotic therapy or causing fever (temperature >100.5°F or 38.1°C) within 1 week prior to first dose.
* Clinically significant other malignancy with the potential to confound study assessments, with the exception of e.g., treated cutaneous squamous cell and basal carcinomas, non-muscle invasive bladder cancer, Rai Stage 0 CLL, and adequately treated Stage 1 to 2 non-cutaneous malignancy in remission for 5 years.
* Subject is unable to comply with the protocol and/or not willing or not available for follow-up assessments
* Subject has any medical intervention or other condition which, in the opinion of the Investigator, could compromise adherence with study requirements or otherwise compromise the study's objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salim Yazji, MD, Study Director — Oncternal Therapeutics
Locations (10):
- United States (9):
  - University of California San Francisco, San Francisco, California
  - Karmanos Cancer Institute, Detroit, Michigan
  - XCancer Omaha, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York
  - NEXT Oncology, Austin, Texas
  - NEXT Oncology, San Antonio, Texas
  - Next Virginia, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- The Royal Marsden NHS Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 40mg QD: 40mg QD of single agent ONCT-534 to be administered daily in oral tablets
  ONCT-534: ONCT-534 is a dual-action androgen receptor inhibitor (DAARI) with a novel mechanism of action that includes inhibition of AR function and degradation of the AR protein mediated by interaction with the N-terminal domain (NTD) of the AR. ONCT-534 has demonstrated preclinical activity in prostate cancer models against both unmutated androgen receptor (AR), and against multiple forms of AR alteration, including those with AR amplification, mutations in the AR ligand binding domain (LBD), and splice variants with loss of the AR LBD.
- Dose Level 2: 80mg QD: 80mg QD of single agent ONCT-534 to be administered daily in oral tablets
  ONCT-534: ONCT-534 is a dual-action androgen receptor inhibitor (DAARI) with a novel mechanism of action that includes inhibition of AR function and degradation of the AR protein mediated by interaction with the N-terminal domain (NTD) of the AR. ONCT-534 has demonstrated preclinical activity in prostate cancer models against both unmutated androgen receptor (AR), and against multiple forms of AR alteration, including those with AR amplification, mutations in the AR ligand binding domain (LBD), and splice variants with loss of the AR LBD.
- Dose Level 3: 160mg QD: 160mg QD of single agent ONCT-534 to be administered daily in oral tablets
  ONCT-534: ONCT-534 is a dual-action androgen receptor inhibitor (DAARI) with a novel mechanism of action that includes inhibition of AR function and degradation of the AR protein mediated by interaction with the N-terminal domain (NTD) of the AR. ONCT-534 has demonstrated preclinical activity in prostate cancer models against both unmutated androgen receptor (AR), and against multiple forms of AR alteration, including those with AR amplification, mutations in the AR ligand binding domain (LBD), and splice variants with loss of the AR LBD.
- Dose Level 4: 300mg QD: 300mg QD of single agent ONCT-534 to be administered daily in oral tablets
  ONCT-534: ONCT-534 is a dual-action androgen receptor inhibitor (DAARI) with a novel mechanism of action that includes inhibition of AR function and degradation of the AR protein mediated by interaction with the N-terminal domain (NTD) of the AR. ONCT-534 has demonstrated preclinical activity in prostate cancer models against both unmutated androgen receptor (AR), and against multiple forms of AR alteration, including those with AR amplification, mutations in the AR ligand binding domain (LBD), and splice variants with loss of the AR LBD.
- Dose Level 5: 600mg QD: 600mg QD of single agent ONCT-534 to be administered daily in oral tablets
  ONCT-534: ONCT-534 is a dual-action androgen receptor inhibitor (DAARI) with a novel mechanism of action that includes inhibition of AR function and degradation of the AR protein mediated by interaction with the N-terminal domain (NTD) of the AR. ONCT-534 has demonstrated preclinical activity in prostate cancer models against both unmutated androgen receptor (AR), and against multiple forms of AR alteration, including those with AR amplification, mutations in the AR ligand binding domain (LBD), and splice variants with loss of the AR LBD.
- Dose Level 6: 1200 mg QD: 1200mg QD of single agent ONCT-534 to be administered daily in oral tablets
  ONCT-534: ONCT-534 is a dual-action androgen receptor inhibitor (DAARI) with a novel mechanism of action that includes inhibition of AR function and degradation of the AR protein mediated by interaction with the N-terminal domain (NTD) of the AR. ONCT-534 has demonstrated preclinical activity in prostate cancer models against both unmutated androgen receptor (AR), and against multiple forms of AR alteration, including those with AR amplification, mutations in the AR ligand binding domain (LBD), and splice variants with loss of the AR LBD.
- BID Dose Level 1: 160 mg BID: 160mg BID of single agent ONCT-534 to be administered daily in oral tablets
  ONCT-534: ONCT-534 is a dual-action androgen receptor inhibitor (DAARI) with a novel mechanism of action that includes inhibition of AR function and degradation of the AR protein mediated by interaction with the N-terminal domain (NTD) of the AR. ONCT-534 has demonstrated preclinical activity in prostate cancer models against both unmutated androgen receptor (AR), and against multiple forms of AR alteration, including those with AR amplification, mutations in the AR ligand binding domain (LBD), and splice variants with loss of the AR LBD.
- BID Dose Level 2: 300 mg BID: 300mg BID of single agent ONCT-534 to be administered twice daily in oral tablets
  ONCT-534: ONCT-534 is a dual-action androgen receptor inhibitor (DAARI) with a novel mechanism of action that includes inhibition of AR function and degradation of the AR protein mediated by interaction with the N-terminal domain (NTD) of the AR. ONCT-534 has demonstrated preclinical activity in prostate cancer models against both unmutated androgen receptor (AR), and against multiple forms of AR alteration, including those with AR amplification, mutations in the AR ligand binding domain (LBD), and splice variants with loss of the AR LBD.
Period: Overall Study
Arm/Group | Dose Level 1: 40mg QD | Dose Level 2: 80mg QD | Dose Level 3: 160mg QD | Dose Level 4: 300mg QD | Dose Level 5: 600mg QD | Dose Level 6: 1200 mg QD | BID Dose Level 1: 160 mg BID | BID Dose Level 2: 300 mg BID
Started | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 3
Safety Population | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 3
DLT-evaluable Pop | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3
Efficacy-evaluable Population | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 3
Not completed — Progressive Disease | 1 | 1 | 2 | 3 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: 40mg QD | Dose Level 2: 80mg QD | Dose Level 3: 160mg QD | Dose Level 4: 300mg QD | Dose Level 5: 600mg QD | Dose Level 6: 1200 mg QD | BID Dose Level 1: 160 mg BID | BID Dose Level 2: 300 mg BID | Total
Number analyzed (Participants) | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 3 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 | 83 | 70.3 (3.0) | 67.3 (4.5) | 70.0 (9.0) | 76.0 (5.6) | 67.7 (11.7) | 74.0 (7.2) | 69.8 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 1 | 4 | 3 | 3 | 3 | 3 | 3 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 1 | 4 | 2 | 3 | 2 | 2 | 3 | 18
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 4 | 3 | 2 | 2 | 3 | 2 | 18
  United Kingdom | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities Through Study Day 28
Description: Incidence of DLTs through Study Day 28
Time Frame: Number of Participants with Dose Limiting Toxicities Through Study Day 28
Population: DLT-evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 40mg QD | Dose Level 2: 80mg QD | Dose Level 3: 160mg QD | Dose Level 4: 300mg QD | Dose Level 5: 600mg QD | Dose Level 6: 1200 mg QD | BID Dose Level 1: 160 mg BID | BID Dose Level 2: 300 mg BID
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Reduction of Prostate-Specific Antigen (PSA) by More Than 50%
Description: Proportion of patients who achieve at least a 50% drop in PSA from baseline (PSA50)
Time Frame: Up to 51 Weeks
Population: Efficacy-evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 40mg QD | Dose Level 2: 80mg QD | Dose Level 3: 160mg QD | Dose Level 4: 300mg QD | Dose Level 5: 600mg QD | Dose Level 6: 1200 mg QD | BID Dose Level 1: 160 mg BID | BID Dose Level 2: 300 mg BID
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Post Hoc Outcome: Number of Subjects With Any Post-Baseline Decrease in PSA
Description: Any reduction in PSA after Baseline (First Day of Treatment)
Time Frame: Up to 51 Weeks
Population: Efficacy-evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 40mg QD | Dose Level 2: 80mg QD | Dose Level 3: 160mg QD | Dose Level 4: 300mg QD | Dose Level 5: 600mg QD | Dose Level 6: 1200 mg QD | BID Dose Level 1: 160 mg BID | BID Dose Level 2: 300 mg BID
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 51 Weeks using the Safety Population
Description: This is based on subjects treated with ONCT-534. 40mg QD (n=1); 80 mg QD (n=1); 160 mg QD (n=4); 300 mg QD (n=3); 600 mg QD (n=3); 1200 mg QD (n=3); 160 mg BID (n=3); 300 mg BID (n=3)
Arm/Group | Dose Level 1: 40mg QD | Dose Level 2: 80mg QD | Dose Level 3: 160mg QD | Dose Level 4: 300mg QD | Dose Level 5: 600mg QD | Dose Level 6: 1200 mg QD | BID Dose Level 1: 160 mg BID | BID Dose Level 2: 300 mg BID
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 1/4 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 2/4 | 1/3 | 1/3 | 2/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 4/4 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: 40mg QD (N=1) | Dose Level 2: 80mg QD (N=1) | Dose Level 3: 160mg QD (N=4) | Dose Level 4: 300mg QD (N=3) | Dose Level 5: 600mg QD (N=3) | Dose Level 6: 1200 mg QD (N=3) | BID Dose Level 1: 160 mg BID (N=3) | BID Dose Level 2: 300 mg BID (N=3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical Haemolytic Uraemic Syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lactic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal Artery Occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: 40mg QD (N=1) | Dose Level 2: 80mg QD (N=1) | Dose Level 3: 160mg QD (N=4) | Dose Level 4: 300mg QD (N=3) | Dose Level 5: 600mg QD (N=3) | Dose Level 6: 1200 mg QD (N=3) | BID Dose Level 1: 160 mg BID (N=3) | BID Dose Level 2: 300 mg BID (N=3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbroscral Plexopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Creatinine Increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extradural Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International Normalised Ratio Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular Block First Degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Creatinine Phophokinase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT05917470/Prot_SAP_003.pdf